CLINICAL TRIAL: NCT01154075
Title: Medication Adherence in Children Who Had a Liver Transplant
Acronym: MALT
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other); University of Pittsburgh (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); University of California, Los Angeles (Other); The Emmes Company, LLC (Industry); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: GCO 09-1112; R01DK080740 (NIH)
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Pediatric Recipients of a Liver Transplant
Keywords: Liver transplant; Adherence; Compliance; Tacrolimus
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — liver tissue samples (from biopsies performed for clinical, not investigational, reasons)
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to evaluate the use of a novel method to measure adherence to immunosuppressant medications in predicting rejection episodes in children who had a liver transplant.

DETAILED DESCRIPTION:
During the course of their illness as many as 50% of children who had a liver transplant stop taking their medications. Non-adherence is the most important reason for organ rejection in long term survivors of pediatric liver transplantation. In order to address this important risk-factor effectively, the first step is to evaluate a method that would identify non-adherence in these children. Medication blood levels that are obtained as a part of clinical practice in transplant centers can be used to determine whether the patient is adherent or not. This multi-center observational study tests the ability of an objective measure of adherence to immunosuppressant medications that involves the use of routinely obtained tacrolimus blood levels to predict organ rejection in children who had a liver transplant.

ELIGIBILITY:
Inclusion Criteria:

* The patient is between > 1 year of age and less than 18 years of age at enrollment
* Guardian's consent, child assent (in accordance with each institution's IRB policies).
* The patient is prescribed tacrolimus (either brand or generic formulation).
* The patient has been seen in the enrolling center's clinic at least once in the last two years.

Exclusion Criteria:

* The patient received a liver transplant less than 1 year prior to enrollment.
* The patient has had more than one solid organ transplant (including marrow replacement).
* The patient has had biopsy-proven rejection within the past six months.
* The patient has been diagnosed with Hepatitis C.
* The guardian or child (in a developmentally-appropriate manner) do not understand the study procedures. This will be verified by asking both guardian and child (if 6 years old or older) to repeat the study procedures.
* The patient is only seen for consultation - most or all of the child's routine care is provided at another center (or in a community clinic).
* Either the patient or the guardian is actively psychotic or severely disoriented due to any cause, including hepatic encephalopathy (temporary exclusion) or severely mentally retarded as defined in the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV).
* The patient is not medically stable or is hospitalized.
* The treating physician has instructed the participant not to obtain tacrolimus levels for at least one year.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients receiving liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 401 (Actual)
Dates: Start 2010-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Rejection episodes | Quarterly for 2 years unless a rejection occurs within this time frame.
  Adherence measured through the use of the standard deviation of a series of tacrolimus blood levels obtained during the course of follow-up is the primary predictor.

SECONDARY OUTCOMES:
Retransplantation or death | 2 years
Liver function tests | Quarterly for 2 years unless a rejection occurs within this time frame.

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Shemesh, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (5):
- United States (5):
  - UCLA Medical Center, Los Angeles, California
  - Children's Memorial Hospital, Chicago, Illinois
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Shemesh E, Bucuvalas JC, Anand R, Mazariegos GV, Alonso EM, Venick RS, Reyes-Mugica M, Annunziato RA, Shneider BL. The Medication Level Variability Index (MLVI) Predicts Poor Liver Transplant Outcomes: A Prospective Multi-Site Study. Am J Transplant. 2017 Oct;17(10):2668-2678. doi: 10.1111/ajt.14276. Epub 2017 Apr 22. PMID 28321975